CLINICAL TRIAL: NCT00327977
Title: A Retrospective Study of Hypoxemia in Infants After Palliative Neonatal Surgery for Congenital Heart Disease
Brief Title: Hypoxemia in Infants After Palliative Surgery
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-128
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: hypoxemia; palliative neonatal surgery
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hypoxia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Congenital heart disease is a major cause of morbidity and mortality in infants. Many cardiac defects require surgical palliation or repair in the newborn period. The effects of chronic hypoxia on growth and development are unclear. Infants with very severe cardiac defects may undergo surgery in infancy, but often this cardiac surgery can provide only palliation, not correction. As a result, these infants are exposed to a physiology of chronic hypoxia during the neonatal period through infancy, a critical period of growth and development. The optimal oxygen saturations for infants with palliated cardiac defects is unknown. The purpose of this study is to analyze the growth and development of infants with post-surgical palliation in infancy and assess variations in oxygenation saturations and hemodynamics as they relate to weight gain, linear growth and increases in head circumference during the first three years of life.

DETAILED DESCRIPTION:
We wish to do a retrospective review of clinical data on infants who have undergone surgical palliation for the following cardiac defects over the past five years (from January 1, 2001 through March 31, 2006):

Hypoplastic left heart syndrome Pulmonary atresia Severe pulmonary stenosis.

The patient charts, between the dates of 01.01.2001and 03.31.2006, will be reviewed from Children's Healthcare of Atlanta, Egleston Hospital and the Sibley Heart Center Cardiology clinics of Children's Healthcare of Atlanta.

We will review approximately 180 charts.

We will collect the following information on each patient:

Medical Record Number Account number Dates of admission, discharge, treatment or death, date of birth Information regarding cardiac signs and symptoms, medication information Age, weight , diagnoses and results of imaging studies Clinic visit information during routine follow up appointments such as weight, length, head circumference, oxygen saturations, vital signs, medications, diet, blood pressures, symptoms,blood tests, chest x-ray findings, dates and types of procedures Readmissions, feeding regimen, cardiac catheterization data, surgical data Parent histories of developmental milestones, physical therapy and speech therapy consultations, feeding history, evaluations of swallowing function Airway symptoms Noncardiac procedures and noncardiac medical problems Family history and social history as it relates to care of the infants at home, complications of medical or surgical treatment and cerebral oximetry.

ELIGIBILITY:
Inclusion Criteria:

* patient charts from 01/01/2001 through 03/31/2006 seen at Children's Healthcare of Atlanta or Sibley Heart Center Cardiology for surgical palliation for Hypoplastic left heart syndrome or surgical palliation for Pulmonary atresia or surgical palliation for Severe pulmonary stenosis

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients'charts only from Children's Healthcare of Atlanta
Sampling Method: Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2001-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Analyze the growth and development of infants with post-surgical palliation in infancy and assess variations in oxygenation saturations and hemodynamics as they relate to weight gain, linear growth and increases in head circumference. | 5 years
  Ongoing data analysis of risk factors for death in the high risk population has revealed that some aspects of the clinical course of these patients which are new to the field. Episodes of decomposition may not have been sudden as previously thought, but may have been preceded by some mild signs of change in cardiovascular status. This may in fact have led to changes in clinical course that were undetected because this was a new clinical finding.

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Clabby, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heart Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States